CLINICAL TRIAL: NCT04345900
Title: A Phase 2, Multicenter, Randomized Study to Evaluate Duration of Severe Neutropenia With Plinabulin Versus Pegfilgrastim in Patients With Solid Tumors Receiving Docetaxel Myelosuppressive Chemotherapy (Protective-1)
Brief Title: Plinabulin vs. Pegfilgrastim in Patients With Solid Tumors Receiving Docetaxel Myelosuppressive Chemotherapy Phase 2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BeyondSpring Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BPI-2358-105 Phase 2
Record Dates: First submitted 2020-03-31; First posted 2020-04-15 (Actual); Results first posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-03

CONDITIONS: Chemotherapy-induced Neutropenia
MeSH Terms: interventions — NPI 2358; pegfilgrastim; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 20 mg/m^2 Plinabulin (Experimental): 75 mg/m^2 Docetaxel + 20 mg/m^2 Plinabulin
  Interventions: Drug: Plinabulin
- 10 mg/m^2 Plinabulin (Experimental): 75 mg/m^2 Docetaxel + 10 mg/m^2 Plinabulin
  Interventions: Drug: Plinabulin
- 5 mg/m^2 Plinabulin (Experimental): 75 mg/m^2 Docetaxel + 5 mg/m^2 Plinabulin
  Interventions: Drug: Plinabulin
- 6 mg Pegfilgrastim (Active Comparator): 75 mg/m^2 Docetaxel + 6 mg Pegfilgrastim
  Interventions: Drug: Pegfilgrastim

INTERVENTIONS:
Drug: Plinabulin — a synthetic, low molecular weight, new chemical entity that belongs to the diketopiperazine class of compounds. Plinabulin is intended for intravenous (IV) infusion and is diluted in D5W and administered for 30 minutes (± 5 minutes).
  Arms: 10 mg/m^2 Plinabulin; 20 mg/m^2 Plinabulin; 5 mg/m^2 Plinabulin
Drug: Pegfilgrastim — PEGFILGRASTIM is a long-acting granulocyte colony-stimulating factor that stimulates the growth of neutrophils, to reduce the incidence of fever and infection in patients with certain types of cancer who are receiving chemotherapy that affects the bone marrow.
  Other Names: G-CSF
  Arms: 6 mg Pegfilgrastim

SUMMARY:
To assess the duration of severe neutropenia (DSN) in treatment Cycle 1 in patients treated with docetaxel (75 mg/m2) + plinabulin (5, 10, or 20 mg/m2) or with docetaxel (75 mg/m2) + pegfilgrastim (6 mg). Neutrophils count was to be assessed at baseline (prior to Cycle 1 docetaxel dose) and during Cycle 1 on Days 1, 2, 6, 7, 8, 9, 10, and 15 (pre-dose on dosing days; times equivalent to pre dose on other days).

DETAILED DESCRIPTION:
55 patients with advanced and metastatic NSCLC have been randomized with the arm designation and planned intervention as follows: Arm 1: Docetaxel (75 mg/m2) + pegfilgrastim (6 mg) Arm 2: Docetaxel (75 mg/m2) + plinabulin (20 mg/m^2) Arm 3: Docetaxel (75 mg/m2) + plinabulin (10 mg/m^2) Arm 4: Docetaxel (75 mg/m2) + plinabulin (5 mg/m^2)

ELIGIBILITY:
Inclusion Criteria:

1. At least ≥ 18 years of age (male or female) at the time of signing the informed consent form.
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
3. Patients with:

   Advanced or metastatic NSCLC failing platinum based therapy
4. Pathology confirmation of cancer
5. Patients with ≥1 of the following risk factors, at the initiation of docetaxel chemotherapy, that would require neutropenia prophylaxis per National Comprehensive Cancer Network (NCCN) guidelines (version 2, 2016) Myeloid Growth Factors:

   1. Prior chemotherapy or radiation treatment
   2. Bone marrow involvement by tumor
   3. Surgery and/or open wounds within 4 weeks of first administration of study drug
   4. Age > 65 years of age and receiving full chemotherapy dose intensity
6. Life expectancy of 3 months or more.
7. The following laboratory results assessed within 14 days prior to study drug administration:

   Hemoglobin ≥ 9 g/dL independent of transfusion or growth factor support ANC ≥ 1.5 x 109/L independent of growth factor support Serum total bilirubin ≤ 1.5 times the upper limit normal (ULN), unless the patient has a diagnosis of Gilbert's disease in which case direct bilirubin ≤ 1.5 times ULN of the direct bilirubin.

   Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN (≤1.5 x ULN if alkaline phosphatase [AP] is > 2.5 x ULN) Serum creatinine ≤ 1.5 x ULN
8. Prothrombin time (PT) and International Normalized Ratio (INR) ≤ 1.5 × upper limit of normal (ULN), activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN, based on central laboratory results.
9. Female patients of childbearing potential who had a negative pregnancy test at screening. Females of childbearing potential are defined as sexually mature women without prior hysterectomy or who have had any evidence of menses in the past 12 months. However, women who have been amenorrhoeic for 12 or more months were still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, anti-estrogens, or ovarian suppression.

Women of childbearing potential (i.e., menstruating women) must have a negative urine pregnancy test (positive urine tests are to be confirmed by serum test) documented within the 24-hour period prior to the first dose of study drug.

Sexually active women of childbearing potential enrolled in the study must agree to use two forms of accepted methods of contraception during the course of the study and for 3 months after their last dose of study drug. Effective birth control includes (a) intrauterine device (IUD) plus one barrier method; (b) on stable doses of hormonal contraception for at least 3 months (e.g., oral, injectable, implant, transdermal) plus one barrier method; (c) 2 barrier methods. Effective barrier methods are male or female condoms, diaphragms, and spermicides (creams or gels that contain a chemical to kill sperm); or (d) a vasectomized partner.

For male patients who were sexually active and who were partners of premenopausal women: agreement to use two forms of contraception during the treatment period and for at least 3 months after the last dose of study drug

Exclusion Criteria:

1. History of myelogenous leukemia, myelodysplastic syndrome or concomitant sickle cell disease.
2. Received chemotherapy within 4 weeks prior to the first dose of study drug.
3. Received prior docetaxel, except adjuvant docetaxel given > 1 year prior to first dose of study drug.
4. Use of strong cytochrome P450 (CYP) 3A4 inhibitors, within 3 days of the first administration of study drug, and 7 days after treatment with taxanes OR required use of strong CYP3A4 inhibitors (refer to Section 10.6.2)
5. Received an investigational agent or tumor vaccine within 2 weeks before the first dose of study drug; patients must have recovered from toxicity of prior treatment and have no > Grade 1 Common Terminology Criteria for Adverse Events (CTCAE) (v4.03) treatment-emergent AEs (TEAEs).
6. Received any concurrent anticancer therapies.
7. Received a prior bone marrow or stem cell transplant.
8. Had a co-existing active infection or received systemic anti-infective treatment within 72 hours before the first dose of study drug.
9. Prior radiation therapy within the 4 weeks before the first dose of study drug.
10. Prior use of pegfilgrastim or filgrastim within 4 weeks before the first dose of study drug.
11. Presence of any serious or uncontrolled illness including, but not limited to: uncontrolled diabetes, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, uncontrolled arterial thrombosis, symptomatic pulmonary embolism, or psychiatric illness that would limit compliance with study requirements, or any other conditions that would preclude the patient from study treatment as per the discretion of the Investigator.
12. Significant cardiovascular history:

    History of myocardial infarction or ischemic heart disease within 1 year (within a window of up to 18 days less than 1 year) before first study drug administration; Uncontrolled arrhythmia; History of congenital QT prolongation; Electrocardiogram (ECG) findings consistent with active ischemic heart disease; New York Heart Association Class III or IV cardiac disease; Uncontrolled hypertension: blood pressure consistently >150 mm Hg systolic and > 100 mm Hg diastolic despite antihypertensive medication.
13. History of hemorrhagic diarrhea, inflammatory bowel disease, or active uncontrolled peptic ulcer disease. (Concomitant therapy with ranitidine or its equivalent and/or omeprazole or its equivalent is acceptable). History of ileus or other significant gastrointestinal disorder known to predispose to ileus or chronic bowel hypomotility.
14. Any other malignancy requiring active therapy.
15. Known human immunodeficiency virus (HIV) seropositivity.
16. Hepatitis B virsu (HBV) or hepatitis C virus (HCV) infection requiring treatment
17. Female subject who is pregnant or lactating.
18. Unwilling or unable to comply with procedures required in this protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2018-03-20 (Actual); Study Completion 2018-04-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- United States (4):
  - Emad Ibrahim, MD, Inc., Redlands, California
  - Mid Florida Hematology & Oncology Center, Orange City, Florida
  - Cancer Center of Middle Georgia, Dublin, Georgia
  - Hematology/Oncology of the North Shore, Skokie, Illinois
- China (3):
  - Harbin Medical University Cancer Hospital, Harbin, Harbin
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
- Russia (3):
  - Medical University 'REAVIZ', Samara
  - SBI of Healthcare "Oncology Dispensary #2" Ministry of Healthcare of Krasnodar Region, Sochi
  - Volgograd Regional Clinical Oncology Dispensary, Volgograd
- Ukraine (9):
  - Municipal Institution Dnipropetrovsk City Multi-functional Hospital, Dnipro
  - Prykarpatian Clinical Oncological Center, Ivano-Frankivsk
  - Kherson regional oncological dispensary Communal Institution of Kherson Regional council, Kherson
  - Regional Municipal Institution "Kryvyy Rig Oncology Dispensary", Krivói Rog
  - Kirovograd Regional Oncological Center, Kropyvnytskyi
  - Kyiv City Clinical Oncology Center, Kyiv
  - Lviv State Oncological Regional Treatment and Preventive Center, Lviv
  - Municipal Institution "Sumy Regional Clinical Oncology Dispensary", Sumy
  - Zakarpattia Regional Clinical Oncology Center, Uzhhorod

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: 75 mg/m^2 Docetaxel + 6 mg Pegfilgrastim
- Arm 2: 75 mg/m^2 Docetaxel + 20 mg/m^2 Plinabulin
- Arm 3: 75 mg/m^2 Docetaxel + 10 mg/m^2 Plinabulin
- Arm 4: 75 mg/m^2 Docetaxel + 5 mg/m^2 Plinabulin
Period: Overall Study
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Started | 13 | 14 | 14 | 14
Completed (l) | 11 | 11 | 10 | 9
Not Completed | 2 | 3 | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Total
Number analyzed (Participants) | 13 | 14 | 14 | 14 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 7 | 9 | 5 | 30
  >=65 years | 4 | 7 | 5 | 9 | 25
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.5 (8.08) | 63.0 (10.44) | 58.6 (11.72) | 64.1 (10.33) | 61.3 (10.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 5 | 5 | 17
  Male | 10 | 10 | 9 | 9 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 4 | 3 | 3 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 10 | 10 | 11 | 11 | 42
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Neutrophil Count at Baseline Visit (Pre-dose) [Mean (Standard Deviation); unit: 10^9 Cells/L] | 9.766 (3.4633) | 7.498 (2.3376) | 8.870 (3.0302) | 8.061 (3.9371) | 8.527 (3.2641)

OUTCOME MEASURES:

1. Primary Outcome: DSN
Description: Duration of Grade 4 neutropenia (ANC < 0.5 × 109/L)
Time Frame: At the end of Cycle 1 (each cycle is 21 days)
Measure: Mean (Standard Deviation); unit: days
Groups:
- Arm 1: 75 mg/m^2 Docetaxel +6 mg Pegfilgrastim
- Arm 2: 75 mg/m^2 Docetaxel +20 mg/m^2 Plinabulin
- Arm 3: 75 mg/m^2 Docetaxel +10 mg/m^2 Plinabulin
- Arm 4: 75 mg/m^2 Docetaxel +5 mg/m^2 Plinabulin
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 13 | 14 | 14 | 14
days | 0.15 (0.376) | 0.36 (0.929) | 0.43 (1.089) | 0.29 (0.611)

2. Secondary Outcome: Peak Plasma Concentration (Cmax)
Description: a parameter to establish the pharmacokinetic profile of plinabulin by evaluating the peak plasma concentration (Cmax) of the drug in the blood after administration of a single dose of the drug
Time Frame: 0, 0.5, 1, 4.5, 24 hours post-dose
Population: Arm 1 is the positive placebo group
Measure: Mean (Standard Deviation); unit: mg/L
Groups:
- Arm 1: 75mg/m^2 Docetaxel + 6 mg Pegfilgrastim
- Arm 2: 75mg/m^2 Docetaxel + 20 mg/m^2 Plinabulin
- Arm 3: 75mg/m^2 Docetaxel + 10 mg/m^2 Plinabulin
- Arm 4: 75mg/m^2 Docetaxel + 5 mg/m^2 Plinabulin
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 0 | 14 | 14 | 14
mg/L |  | 0.263 (0.173) | 0.131 (0.086) | 0.066 (0.043)

3. Secondary Outcome: Area Under Curve (AUC)
Description: A parameter to establish the pharmacokinetic profile of plinabulin to describe the variation of the drug concentration in blood plasma as a function of time
Time Frame: 0, 0.5, 1, 4.5, 24 hours post-dose
Population: Arm 1 is positive placebo group
Measure: Median (Standard Deviation); unit: mg*hr/L
Groups:
- Arm2: 75 mg/m^2 Docetaxel +20 mg/m^2 Plinabulin
Arm/Group | Arm 1 | Arm2 | Arm 3 | Arm 4
Number analyzed (Participants) | 0 | 14 | 14 | 14
mg*hr/L |  | 1.22 (1.56) | 0.61 (0.78) | 0.31 (0.39)

4. Secondary Outcome: Terminal Half-time (T1/2)
Description: A parameter to establish the pharmacokinetic profile of plinabulin by measuring the time it takes for the concentration of the drug in the plasma to be reduced by 50%
Time Frame: 0, 0.5, 1, 4.5, 24 hours post-dose
Population: Arm 1 is positive placebo group
Measure: Median (Standard Deviation); unit: hrs
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 0 | 14 | 14 | 14
hrs |  | 7.38 (3.26) | 7.39 (1.79) | 7.99 (3.69)

5. Secondary Outcome: Volume of Distribution in the Terminal Elimination Phase (Vz)
Description: A parameter to establish the pharmacokinetic profile of plinabulin by evaluating Vz.
Time Frame: 0, 0.5, 1, 4.5, 24 hours post-dose
Population: Arm 1 is the positive placebo group
Measure: Median (Standard Deviation); unit: L
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 0 | 14 | 14 | 14
L |  | 198 (51) | 248 (72) | 154 (111)

6. Secondary Outcome: Clearance (Cl)
Description: a parameter to establish the pharmacokinetic profile of plinabulin
Time Frame: 0, 0.5, 1, 4.5, 24 hours post-dose
Population: Arm 1 is positive Placebo group
Measure: Median (Standard Deviation); unit: L/hr
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 0 | 14 | 14 | 14
L/hr |  | 22.9 (18.0) | 25.0 (15.0) | 18.5 (23.7)

7. Secondary Outcome: Systolic Blood Pressure
Description: a parameter to establish the pharmacodynamic profile of plinabulin
Time Frame: 0, 0.5, 1, 4.5, 24 hours post-dose
Population: Arm 1 is the positive placebo group
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 0 | 14 | 14 | 14
mm Hg |  | 136 (24) | 134 (18.7) | 138 (19.5)

8. Secondary Outcome: Diastolic Blood Pressure
Description: a parameter to establish the pharmacodynamic profile of plinabulin
Time Frame: 0, 0.5, 1, 4.5, 24 hours post-dose
Population: Arm 1 is positive placebo group
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 0 | 14 | 14 | 14
mm Hg |  | 79.2 (11.6) | 84.1 (16.8) | 84.8 (13.0)

9. Secondary Outcome: Area Over the Neutropenia Curve
Description: a parameter to establish the pharmacodynamic profile of plinabulin
Time Frame: 0, 0.5, 1, 4.5, 24 hours post-dose
Population: Arm 1 is positive placebo group
Measure: Mean (Standard Deviation); unit: mg*hr/L
Arm/Group | Arm 1 | Arm2 | Arm 3 | Arm 4
Number analyzed (Participants) | 0 | 14 | 14 | 14
mg*hr/L |  | 0.086 (0.815) | 0.111 (0.955) | 0.113 (0.958)

ADVERSE EVENTS:
Time Frame: Time of screening until 30 day follow up (5 months).
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
All-Cause Mortality (participants affected / at risk) | 1/13 | 1/14 | 1/14 | 1/14
Serious Adverse Events (participants affected / at risk) | 2/13 | 2/14 | 2/14 | 2/14
Other Adverse Events (participants affected / at risk) | 11/13 | 12/14 | 12/14 | 12/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (N=13) | Arm 2 (N=14) | Arm 3 (N=14) | Arm 4 (N=14)
Atrial Fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Vomitting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0
Disease Progression (General disorders) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Septic Shock (Infections and infestations) | 0 | 1 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (N=13) | Arm 2 (N=14) | Arm 3 (N=14) | Arm 4 (N=14)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 5 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Haemorrhagic Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 4 | 5 | 6 | 7
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 3
Neutropenia (Blood and lymphatic system disorders) | 3 | 7 | 5 | 9
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac Failure (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial Firbrosis (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial Ischaemia (Cardiac disorders) | 1 | 0 | 0 | 0
Sinus Tachycardia (Cardiac disorders) | 2 | 0 | 1 | 0
Supraventricular Extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 1
Tachycardia (Cardiac disorders) | 2 | 0 | 0 | 0
Chalazion (Eye disorders) | 0 | 1 | 0 | 0
Dry Eye (Eye disorders) | 0 | 0 | 0 | 1
Mydriasis (Eye disorders) | 0 | 0 | 0 | 1
Abdominal Distension (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Anal Incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 1 | 4
Nausea (Gastrointestinal disorders) | 2 | 2 | 0 | 2
Oral Mucosal Blistering (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Regurgitation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Retching (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Vomitting (Gastrointestinal disorders) | 0 | 2 | 0 | 2
Asthenia (General disorders) | 0 | 1 | 0 | 1
Chest Discomfort (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 1 | 3 | 4
Gait Disturbance (General disorders) | 0 | 0 | 0 | 1
Localized Oedema (General disorders) | 0 | 0 | 0 | 1
Mucosal Inflammation (General disorders) | 0 | 0 | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 1 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 1
Odema Peripheral (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1 | 1
Liver Injury (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Angular Cheilitis (Infections and infestations) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Respiratory Tract Infection Viral (Infections and infestations) | 1 | 0 | 1 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1
Viral Infection (Infections and infestations) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Foot Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Alanine Aminotransferase increased (Investigations) | 0 | 0 | 1 | 1
Amylase Increased (Investigations) | 0 | 1 | 0 | 0
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 2 | 0
Blood Bilirubin Increased (Investigations) | 0 | 0 | 1 | 0
Blood Creatinine Increased (Investigations) | 0 | 0 | 1 | 0
Blood Glucose Increased (Investigations) | 1 | 0 | 0 | 0
Blood Pressure Increased (Infections and infestations) | 0 | 0 | 0 | 1
Grip Strength Decreased (Investigations) | 0 | 0 | 0 | 1
Neutrophil Count Decreased (Investigations) | 0 | 1 | 2 | 0
Platelet Count Decreased (Investigations) | 0 | 0 | 1 | 0
Weight Decreased (Investigations) | 0 | 1 | 0 | 0
White Blood Cell Count Decreased (Investigations) | 1 | 1 | 3 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 1 | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Complex Regional Pain Syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Hypogeusia (Nervous system disorders) | 0 | 0 | 1 | 0
Neuropathy Peripheral (Nervous system disorders) | 1 | 1 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1
Mood Altered (Psychiatric disorders) | 0 | 1 | 0 | 0
Urinary Incontinence (Psychiatric disorders) | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Chronic Obstructive Pulmonry Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 4 | 7 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Haemorrhage Subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Nail Disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin Discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin Disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Flushing (Vascular disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 4 | 2
Hypotension (Vascular disorders) | 0 | 1 | 0 | 1
Superior Vena Cava Syndrome (Vascular disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-05-30): https://cdn.clinicaltrials.gov/large-docs/00/NCT04345900/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-07): https://cdn.clinicaltrials.gov/large-docs/00/NCT04345900/SAP_001.pdf